CLINICAL TRIAL: NCT05236647
Title: The SIM-study: A Randomized Controlled Trial of Subcutaneous Versus Intravenous Morphine When Switching From Oral to Parenteral Route in Palliative Cancer Patients
Brief Title: Subcutaneous Versus Intravenous Morphine When Switching From Oral to Parenteral Route in Palliative Cancer Patients
Acronym: SIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Olav Fredheim, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/291056(REK)
Record Dates: First submitted 2022-01-26; First posted 2022-02-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Pain Cancer
MeSH Terms: conditions — Cancer Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous morphine infusion (Experimental): Morphine 10 mg/ml or morphine 20 mg/ml will be diluted with normal saline to 5 mg/ml or 10 mg/ml. Both active study medication and placebo will be prepared in 100 ml drug containers suitable for the infusion pump.
  The patient will have two similar infusion pumps. Morphine infusion connected to an i.v. line, placebo (normal saline) connected to a s.c line. Bolus dose will initially be equal to dose/hour. The nurse will administer bolus doses on both pumps (placebo and morphine pump) simultaneously. Patient reported pain intensity (NRS 0-10) and whether the bolus dose was initiated by the patient or the nurse will be recorded before each bolus dose. Bolus dose will be equally increased if/when the infusion rate is increased. If the bolus dose is ineffective, the bolus dose can be increased in steps of 0.1 ml until an effective dose is reached.
  Interventions: Drug: Morphine
- Subcutaneous morphine infusion (Active Comparator): Morphine 10mg/ml or morphine 20 mg/ml will be diluted with normal saline to 5 mg/ml or 10 mg/ml. Both active study medication and placebo will be prepared in 100 ml drug containers suitable for the infusion pump.
  The patient will have two similar infusion pumps. Morphine infusion connected to a s.c. line, placebo (normal saline) connected to a i.v. line. Bolus dose will initially be equal to dose/hour. The nurse will administer bolus doses on both pumps (placebo and morphine pump) simultaneously. Patient reported pain intensity (NRS 0-10) and whether the bolus dose was initiated by the patient or the nurse will be recorded before each bolus dose. Bolus dose will be equally increased if/when the infusion rate is increased. If the bolus dose is ineffective, the bolus dose can be increased in steps of 0.1 ml until an effective dose is reached.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Intravenous morphine infusion compared to subcutaneous morphine infusion
  Other Names: Morphine hydrochloride trihydrate

SUMMARY:
The investigators aim to establish whether the intravenous or the subcutaneous route of administration has clinically significant advantages when parenteral administration of morphine is started with a combination of continuous infusion and bolus doses in palliative cancer patients.

Patients admitted to a Hospital palliative medicine unit with an indication for parenteral administration of morphine will be recruited.

The patients will have two similar infusion pumps with continuous infusion and bolus function. One infusion pump will be connected to an intravenous line, the other to a subcutaneous line. One pump contains morphine, one placebo. The primary endpoint is the time from initiation of infusion with titration to the final infusion rate that provides pain control is reached.

DETAILED DESCRIPTION:
Intravenous administration has theoretical advantages in more predictable pharmacokinetics and shorter time to maximum effect. Subcutaneous administration is less invasive, requires less specialized personnel and equipment, and probably poses a lower risk of complications than an intravenous line. Traditionally the subcutaneous route has been the recommended first choice for parenteral administration of opioids for palliative cancer patients.

The investigators aim to establish whether the intravenous or the subcutaneous route of administration has clinically significant advantages when parenteral administration of morphine is started with a combination of continuous infusion and bolus doses in palliative cancer patients.

Patients admitted to a Hospital palliative medicine unit with an indication for parenteral administration of morphine will be recruited.

The patients will have two similar infusion pumps with continuous infusion and bolus function. One infusion pump will be connected to an intravenous line, the other to a subcutaneous line. One pump contains morphine, one placebo. The primary endpoint is the time from initiation of infusion with titration to the final infusion rate that provides pain control is reached. Secondary endpoints are time from bolus administration to pain relief, comparison of Tmax, Cmax, and size of AUC0-60 after bolus doses, the number of bolus doses first 24 and 48 hours, and the number of patients reaching acceptable pain relief within 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Unsatisfactory pain control despite titration of oral or transdermal opioids
* Planned discharge to home or nursing home

Exclusion Criteria:

* Estimated survival time <2 weeks
* A clear indication for either intravenous or subcutaneous administration
* Patient unable to report patient reported outcomes needed in the study due to language barriers or cognitive impairment
* Impossible to establish venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Time from initiation of i.v./s.c. morphine to stable infusion rate is reached | 48 hours
  Time from initiation of i.v./s.c. morphine to stable infusion rate is reached

SECONDARY OUTCOMES:
Number of patients not reaching adequate pain relief. | 48 hours
  Number of patients in each arm not reaching adequate pain relief within 48 hours.
Number of bolus doses first 24 hours and 48 hours | 24 and 48 hours
  Total number of bolus doses first 24 hours and 48 hours
Time from bolus administration to clinically significant pain relief | 60 minutes
  Time from bolus administration to a reduction of minimum 2 on a 0-10 numeric rating scale.
Time to maximum plasma concentration (Tmax). | 120 minutes
  Time to maximum plasma concentration (Tmax) after bolus dose of morphine.
Maximum plasma concentration (Cmax). | 120 minutes
  Maximum plasma concentration (Cmax) after bolus dose of morphine
Area under the plasma concentration versus time curve (AUC). | 120 minutes
  Area under the plasma concentration versus time curve (AUC) after bolus administration of morphine.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Fredheim, MD PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT05236647/SAP_000.pdf